CLINICAL TRIAL: NCT07233811
Title: DARSH - A Multicenter Randomized Controlled Trial: Day-care vs Overnight Stay in Robotic Assisted Hysterectomy in Patients With Bening Disease and Endometrial Cancer.
Brief Title: Day Care in Robotic Surgery Hysterectomy. Investigate Quality of Life and Safety With Same Day Discharge After Robotic Hysterectomy for Patients With Benign and Malignant Disease. A Multicenter Randomized Study With 3 Hospitals in Stockholm Sweden.
Acronym: DARSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Malin Brunes, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-05648-01
Record Dates: First submitted 2025-10-02; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hysterectomy; Same Day Discharge; Robotic Surgical Procedures
Keywords: Hysterectomy; Same day discharge; Robotic assisted Hysterectomy; Robotic suregery
MeSH Terms: interventions — Day Care, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day care (Experimental): The patient returns to home the same day as the surgery is performed (before midnight)
  Interventions: Other: Day care
- Overnight stay (Active Comparator): The patient stay at the hospital overnight after their surgery.
  Interventions: Other: Overnight stay

INTERVENTIONS:
Other: Day care — The patient return to home the same day as the surgery is performed.
  Arms: Day care
Other: Overnight stay — The patient spend the night at the hospital and can not go home until the next morning.
  Arms: Overnight stay

SUMMARY:
Patients undergoing robotic assisted hysterectomy in three different hospitals in Stockholm will be randomized to day-care (going home the same day as the surgery) or admission (staying at least one night after surgery). The aim with this study is to investigate if patients in day-care recover as fast/faster as the other group that stays in the hospital. Both patients with benign disease and malign disease (endometrial cancer) will be included in the study.

Patients quality of life (QoL) will be measured before surgery and after surgery at day 3,7 and 30 with a questionnaire called Eq-5D-5L from Euroqol. The questionnaire is validated for postoperative QoL and widely used.

Complications due to surgery within the 30 first days after surgery will also be recorded in the two groups to make sure it is safe for the patients to go home the same day as their surgery.

DETAILED DESCRIPTION:
The study is a multicenter randomized non-inferiority trial. Three hospitals will participate in the study, Södersjukhuset and Danderyds sjukhus for benign indications, and Karolinska Sjukhuset Solna in case of endometrial cancer. The experimental group consisting of patients undergoing same-day discharge, while the control group consisting of patients admitted overnight. The study will use a 1:1 randomization ratio between the experimental and the control group with stratification for malignant and benign cases, given that Karolinska University Hospital Solna only handles endometrial cancer cases, while the other two sites handle benign cases exclusively.

To measure Quality of Life, the validated Euroqol instrument EQ-5D-5L will be used. The EQ-5D-5L instrument is well validated and used in several studies. The literature support that a 5 points difference at the visaul analog scale (VAS) scale is significant for better/worse health QoL.

To measure patient satisfaction with the length of hospital stay and care given they will at day 30 receive an additional questionnaire, the "Quality in patent perspective" (QPP), which is a validated questionnaire in Swedish.

ELIGIBILITY:
Inclusion Criteria:

* Patient that are planned to undergo total robotic hysterectomy with or without adnexal surgery at the three sites.
* Both benign conditions and endometrial cancer.
* All BMI groups and all uterus sizes.

Exclusion Criteria:

* Age not over 75 years old,
* No company at home first night after surgery
* ASA class 3 that is not only because of high BMI.
* Simultaneous prolapse surgery/lymph node evacuation.
* Severe endometriosis or patients with chronic pain conditions that have a special pain regimen after surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only people with uterus undergoing a hysterectomy can participate in the study.
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QoL) day 3 after surgery compared to before surgery | 3 days
  Patients self reported quality of life (QoL) at a visual analog scale (VAS-scale) as reported in the 5-level EQ-5D Euroqol form (Eq-5d-5L) before surgery, compared with day 3 after surgery. The VAS-Scale goes from 0 to 100 where 0 i labeled "The worst health you can imagine" and 100 is labeled "The best health you can imagine". Compared between the two groups: day care and overnight stay.

SECONDARY OUTCOMES:
Quality of life (QoL) day 30 after surgery. | 30 days
  The patients self-reported value at the VAS-Scale (0-100) as reported in the EQ-5D-5L questionnaire at day 30 compared to their value before surgery.
Patient satisfaction with length of stay | 30 days
  Patient satisfaction with length of stay from the QPP (quality from patients perspective) questionnaire after 30 days.
Eq5D-5L index value of QoL. | 30 days
  The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. These five questions generate an index value ranging from -0,59 to 1, where 1 signifies excellent health and below 0 is worse than death.
Complications after surgery | 30 days
  Complications within 30 days from surgery according to Clavien-Dindo (grouped as None, Grade 1-2, Grade 3 or Grade 4).
Readmission | 30 days
  Readmission to the hospital within 30 days (yes/no
Reoperation | 30 days
  Reoperation within 30 days (yes/no)
Sick leave after suregery | 60 days.
  Length of sick leave after operation, information from the Swedish Social insurance system.
Socioeconomic costs | 30 days
  Socioeconomic cost, "Quality-adjusted life years" (QALY´s). The cost is calculated from the patients Eq5D-5L ratio combined with sick leave and costs for the surgery and care at hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Brunes, MD,PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Södersjukhuset, Stockholm
  - Danderyd Hospital, Stockholm
  - Karolinska University hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data that underlie the reported results.
Supporting Information: SAP, ICF
Time Frame: Beginning 9 month following article publication. Ending 36 month after publication.
Access Criteria: Researchers that provides a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee. A data-sharing agreement will be required. contact: malin.brunes@regionstockholm.se